CLINICAL TRIAL: NCT04408430
Title: The Safety and Effectiveness of the Edwards SAPIEN 3, SAPIEN 3 Ultra, and SAPIEN 3 Ultra RESILIA (SAPIEN 3/Ultra/RESILIA) Valve in Patients With Symptomatic Severe Calcific Mitral Valve Disease With Severe Mitral Annular Calcification Who Are Not Candidates for Standard Mitral Valve Surgery.
Brief Title: The MITRAL II Pivotal Trial (Mitral Implantation of TRAnscatheter vaLves).
Acronym: MITRAL-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayra Guerrero (Other)
Responsible Party: Sponsor-Investigator, Mayra Guerrero, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-002438
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Mitral Annular Calcification; Mitral Stenosis; Mitral Regurgitation; Mitral Valve Disease
Keywords: Transcatheter Mitral Valve Replacement
MeSH Terms: conditions — Mitral Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: 210 subjects: 110 in treatment arm and 100 in registry of medical treatment for patients who are not eligible for treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transseptal ViMAC (Experimental): 110 MAC patients treated with transseptal Valve-in-MAC.
  Interventions: Device: Transseptal ViMAC
- Registry of untreated patients (No Intervention): 100 MAC patients not eligible for transseptal ViMAC, treated with conservative management including medications.

INTERVENTIONS:
Device: Transseptal ViMAC — Transseptal TMVR using balloon-expandable aortic transcatheter valves.
  Other Names: ViMAC
  Arms: Transseptal ViMAC

SUMMARY:
A prospective multicenter study enrolling high surgical risk patients with severe mitral annular calcification (MAC) and symptomatic mitral valve dysfunction (severe stenosis, ≥ moderate to severe regurgitation, or mixed ≥ moderate stenosis and ≥ regurgitation). There are 2 Arms in this study: 1) "Transseptal (TS) Valve-in-MAC" (ViMAC) Arm, and 2) Natural History of Disease Registry (NHDR) for patients treated with medical treatment only (which includes patients who meet inclusion criteria but can't be treated with transeptal ViMAC due to the presence of anatomical exclusion criteria or other exclusion criteria) and have not had other procedures that may impact outcomes (i.e., alcohol septal ablation or radiofrequency ablation). The study also includes a Registry of Permanently Unassigned" for subjects who undergo preemptive septal ablation procedures (alcohol or radiofrequency) in anticipation of continuing onto ViMAC arm, but are not accepted in the ViMAC Study arm or the patient chooses not to undergo ViMAC procedure.

DETAILED DESCRIPTION:
STUDY OBJECTIVE

The purpose of this study is to establish the safety and effectiveness of the Edwards SAPIEN 3, SAPIEN 3 Ultra and SAPIEN 3 Ultra RESILIA (SAPIEN 3/Ultra/RESILIA) valves with Commander delivery system in patients with severe mitral annular calcification and symptomatic mitral valve dysfunction who are not candidates for standard mitral valve surgery.

STUDY DESIGN

A prospective multicenter study enrolling high surgical risk patients with severe mitral annular calcification (MAC) and symptomatic mitral valve dysfunction (severe stenosis, ≥ moderate to severe regurgitation, or mixed ≥ moderate stenosis and ≥ regurgitation). There are 2 arms in this study: 1) "Transseptal (TS) Valve-in-MAC (ViMAC)" arm, 2) Natural History of Disease Registry (NHDR). Patients treated with medical treatment only (which will include patients who meet inclusion criteria but can't be treated with transseptal ViMAC due to the presence of anatomical exclusion criteria or other exclusion criteria) and have not had other procedures that may impact outcomes (i.e. alcohol septal ablation, radiofrequency ablation).

Enrollment Enrollment will consist of 110 patients in the treatment arm (transseptal ViMAC) and up to 100 in the medically treated arm).

ELIGIBILITY:
Inclusion Criteria:

All Candidates must meet the following criteria:

1. - 18 years of age or older
2. -Severe mitral annular calcification with symptomatic mitral valve dysfunction including severe mitral stenosis defined as mitral valve area (MVA) of ≤1.5 cm2, or ≥ moderate to severe mitral regurgitation, or mixed ≥ moderated stenosis and ≥ moderate regurgitation. For this study, the severity of mitral regurgitation will be graded according to the 2017 American Society of Echocardiography Guidelines: None, Trivial, Mild 1(+), Moderate 2(+), Moderate to severe 3(+), and severe 4(+).
3. - NYHA Functional Class ≥II.
4. The heart team agrees that valve implantation will likely benefit the patient.
5. High or prohibitive risk for standard mitral valve surgery as determined by the heart team (at least one site cardiac surgeon must personally examine the subject to determine operative risk in patients presented for inclusion to ViMAC arm). NOTE: Patients not interested in mitral intervention or who are being considered for inclusion in the Natural History of Disease Registry are not required to be evaluated in person by a surgeon.)
6. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
7. The study patient agrees to comply with all required post-procedure follow-up visits including annual visits through 5 years.

Exclusion Criteria for ViMAC subjects (does not apply to the Natural History of Disease Registry):

1. - The heart team considers the patient is a surgical candidate.
2. - Mitral annulus is not severely calcified.
3. - Myocardial infarction requiring revascularization within 30 days from procedure.
4. - Clinically significant untreated coronary artery disease requiring revascularization.
5. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease). Implantation of a permanent pacemaker is not exclusionary.
6. Any patient with a balloon valvuloplasty (BMV) within 30 days of the procedure (unless BMV is a bridge to ViMAC procedure after a qualifying Echo).
7. Severe symptomatic tricuspid regurgitation (hepatic dysfunction, ascites, edema not controlled with diuretics) requiring surgery.
8. Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb < 9 g/dL), Thrombocytopenia (Platelets < 50,000 cell/mL), history of coagulopathy or hypercoagulable state.
9. Hypertrophic obstructive cardiomyopathy (HOCM) with mean LVOT gradient of ≥20 mm Hg at rest or ≥50 mmHg with Valsalva.
10. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of screening evaluation.
11. Need for emergency surgery for any reason.
12. Severe left ventricular dysfunction with LVEF < 20%.
13. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
14. Active upper GI bleeding within 90 days prior to procedure.
15. A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure.
16. Cardiac anatomy that would preclude appropriate delivery and deployment of an Edwards SAPIEN 3/Ultra/RESILIA valve in MAC via transseptal access, including but not limited to:

    * Native neo mitral annulus size < 275 mm2 or > 810 mm2 as measured by CT scan.
    * Significant risk of LVOT obstruction or valve embolization as assessed by CT core lab
17. Clinically (by neurologist) or neuroimaging confirmed stroke or transient ischemic attack (TIA) within 90 days of the procedure.
18. Estimated life expectancy <12 months due to non-cardiac conditions.
19. Expectation that patient will not improve despite treatment of mitral valve dysfunction.
20. Active bacterial endocarditis within 180 days of procedure.
21. - Severe right ventricular dysfunction as assessed by Echo core lab
22. - Active infection requiring antibiotic therapy (subject may be a candidate after 2 weeks of antibiotic discontinuation.
23. - Female who is pregnant or lactating.
24. - Participating in another investigational device study.
25. - Aortic valve disease requiring intervention. If aortic valve intervention is required, the AVR procedure should be performed first and if the patient remains symptomatic after AVR, may be presented for consideration for inclusion in this trial.
26. - Severe fixed pulmonary hypertension (PASP ≥70 mmHg and more than 2/3 of the systemic systolic blood pressure).
27. - Severe chronic obstructive pulmonary disease requiring continuous home oxygen.
28. - The patient refuses mitral valve intervention
29. - Recent symptomatic COVID-19 infection with residual symptoms that may affect the outcomes of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: All Cause Morality and Hospitalization for Heart Failure | 1 year.
  A non-hierarchical composite of all-cause mortality and hospitalization for heart failure.

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint | 1 year
  • Stroke at 30 days and 1 year.
Secondary Effectiveness Endpoint | 1 year.
  • Change from baseline in New York Heart Association Class at 1 year.
Secondary Effectiveness Endpoint | 1 year.
  • Change from baseline in distance walked measure by the 6 Minute Walk Test at 1 year.
Secondary Effectiveness Endpoint | 1 year.
  • Change from baseline in quality-of-life measure by the Kansas City Cardiomyopathy Questionnaire (KCCQ) at 1 year.
Secondary Effectiveness Endpoint | 1 year.
  • Echocardiographic assessment of degree of mitral regurgitation (central and paravalvular) at 1 year.
Secondary Effectiveness Endpoint | 1 year.
  • Significant mitral stenosis defined as mean mitral valve gradient by echo > 10 mmHg at 1 year.

OTHER OUTCOMES:
Additional Endpoint: Technical Success | Immediately after the intervention procedure.
  • Technical success at exit from the cath lab.
  Defined as:
  * Successful vascular access, delivery and retrieval of the transcatheter valve delivery system.
  * Deployment of a single valve.
  * Correct position of transcatheter valve in the mitral annulus.
  * Adequate performance of the prosthetic heart valve (MVA > 1.5 cm2) without residual mitral regurgitation grade ≥2 (+).
  * No need for additional surgery or re-intervention (includes drainage of pericardial effusion).
  * The patient leaves the cath lab alive.
Additional Endpoint: Procedural Success | 30 days
  • Procedural Success at 30 days.
  Defined as:
  * Device success at 30 days.
  * No device/procedure related SAE's including: death, stroke, MI or coronary ischemia requiring PCI or CABG, stage 2 or 3 AKI including dialysis, life threatening bleeding, major vascular or access complications (arterial, venous, or TA - any event requiring additional unplanned surgical or transcatheter intervention), pericardial effusion or tamponade requiring drainage, severe hypotension, heart failure or respiratory failure requiring intravenous pressors or invasive or mechanical treatments such as ultrafiltration or hemodynamic assist devices including intra-aortic balloon pump or left ventricular assist device, or prolonged intubation for ≥48 hrs, or any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention.
Additional Endpoint: Device Success | 30 days.
  Device success is defined as:
  * Stroke free survival with original valve in place.
  * No need for additional surgery or re-intervention related to the procedure, access or to the replacement valve.
  * Proper placement and intended function of the replacement valve, including
  * No migration, fracture, thrombosis, hemolysis or endocarditis.
  * No replacement valve stenosis (MV gradient < 10 mmHg).
  * Replacement valve regurgitation < 2 + (including central and paravalvular leak) and without associated hemolysis.
  * No increase in AI from baseline (more than 1 grade) and LVOT gradient < 20 mmHg increase from baseline.
Additional Efficacy Endpoint - NYHA Class at 30 days. | 30 days.
  • Change from baseline in NYHA Class at 30 days.
Additional Efficacy Endpoint - Distance walked in 6 MWT at 30 days | 30 days.
  • Change from baseline in distance walked measure by the 6 MWT at 30 days.
Additional Efficacy Endpoint - KCCQ at 30 days | 30 days.
  • Change from baseline in KCCQ at 30 days.
Additional Efficacy Endpoint - MR severity at 30 days | 30 days
  • Degree of mitral regurgitation (central and paravalvular) at 30 days.
Additional Safety Endpoint - Stroke at 30 days and 1 year. | 30 days and 1 year.
  • Stroke at 30 days and 1 year.
Additional Safety Endpoint - Need for ASD Closure | 30 days.
  • Iatrogenic ASD causing RV failure or hypoxemia or need for ASD closure at discharge and 30 days.
Additional Safety Endpoint - New LVOT Gradient | 30 days and 1 year.
  • New mean LVOT gradient ≥ 20 mmHg, or ≥ 20 mmHg increase from baseline LVOT gradient at 30 days and 1 year.
Additional Efficacy Endpoint - Mitral Valve Reintervention | 30 days and 1 year.
  • Mitral Valve reintervention at 30 days and 1 year.
Additional Safety Endpoint - Hospitalizations at 1 year | 1 year.
  • Number of hospitalizations at 1 year.
Additional Efficacy Endpoint - Days Alive Out of the Hospital | 1 year.
  • Days alive out of hospital at 1 year from index procedure (ViMAC arm) or from assignment day (Natural History Registry).
Additional Safety Endpoint - Hemolysis | 30 days and 1 year.
  • Hemolysis at 30 days and 1 year.
Additional Safety Endpoint - Endocarditis | 30 days and 1 year.
  • Endocarditis at 30 days and 1 year.
Additional Safety Endpoint - Blood Transfusion | 30 days and 1 year.
  • Blood transfusion at 30 days and 1 year.
Additional Safety Endpoint - New Pacemaker Requirement | 30 days and 1 year.
  • New pacemaker requirement at 30 days and 1 year.
Additional Safety Endpoint - New Aortic Valve Insufficiency | 30 days and 1 year.
  • New aortic valve insufficiency at 30 days and 1 year.
Additional Safety Endpoint - Acute Kidney Injury | 30 days and 1 year.
  • Acute kidney injury (MVARC) at 30 days and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mayra Guerrero, MD, Principal Investigator — Mayo Clinic
Locations (17):
- United States (16):
  - Dignity Health Chandler Regional Medical Center, Gilbert, Arizona
  - Banner - University Medicine Cardiology Clinic, Phoenix, Arizona
  - Pima Heart & Vascular, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Health, San Francisco, California
  - Uchealth Heart & Vascular Clinic Harmony Campus, Fort Collins, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center/NYPH, New York, New York
  - Oklahoma Heart Institute Utica Office, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University Health, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - The Sentara Heart Valve and Structural Disease Center, Norfolk, Virginia
- Ignacio Chávez National Institute of Cardiology, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russell HM, Guerrero ME, Salinger MH, Manzuk MA, Pursnani AK, Wang D, Nemeh H, Sakhuja R, Melnitchouk S, Pershad A, Fang HK, Said SM, Kauten J, Tang GHL, Aldea G, Feldman TE, Bapat VN, George IM. Open Atrial Transcatheter Mitral Valve Replacement in Patients With Mitral Annular Calcification. J Am Coll Cardiol. 2018 Sep 25;72(13):1437-1448. doi: 10.1016/j.jacc.2018.07.033. PMID 30236304
- [Background] Guerrero M, Wang DD, Himbert D, Urena M, Pursnani A, Kaddissi G, Iyer V, Salinger M, Chakravarty T, Greenbaum A, Makkar R, Vahanian A, Feldman T, O'Neill W. Short-term results of alcohol septal ablation as a bail-out strategy to treat severe left ventricular outflow tract obstruction after transcatheter mitral valve replacement in patients with severe mitral annular calcification. Catheter Cardiovasc Interv. 2017 Dec 1;90(7):1220-1226. doi: 10.1002/ccd.26975. Epub 2017 Mar 7. PMID 28266162
- [Background] Guerrero M, Wang DD, O'Neill W. Percutaneous alcohol septal ablation to acutely reduce left ventricular outflow tract obstruction induced by transcatheter mitral valve replacement. Catheter Cardiovasc Interv. 2016 Nov 15;88(6):E191-E197. doi: 10.1002/ccd.26649. Epub 2016 Jul 5. PMID 27377756
- [Background] Guerrero M, Urena M, Pursnani A, Wang DD, Vahanian A, O'Neill W, Feldman T, Himbert D. Balloon expandable transcatheter heart valves for native mitral valve disease with severe mitral annular calcification. J Cardiovasc Surg (Torino). 2016 Jun;57(3):401-9. PMID 27094423
- [Background] Guerrero M, Greenbaum A, O'Neill W. First in human percutaneous implantation of a balloon expandable transcatheter heart valve in a severely stenosed native mitral valve. Catheter Cardiovasc Interv. 2014 Jun 1;83(7):E287-91. doi: 10.1002/ccd.25441. Epub 2014 Mar 14. PMID 24532349
- [Result] Guerrero M, Urena M, Himbert D, Wang DD, Eleid M, Kodali S, George I, Chakravarty T, Mathur M, Holzhey D, Pershad A, Fang HK, O'Hair D, Jones N, Mahadevan VS, Dumonteil N, Rodes-Cabau J, Piazza N, Ferrari E, Ciaburri D, Nejjari M, DeLago A, Sorajja P, Zahr F, Rajagopal V, Whisenant B, Shah PB, Sinning JM, Witkowski A, Eltchaninoff H, Dvir D, Martin B, Attizzani GF, Gaia D, Nunes NSV, Fassa AA, Kerendi F, Pavlides G, Iyer V, Kaddissi G, Witzke C, Wudel J, Mishkel G, Raybuck B, Wang C, Waksman R, Palacios I, Cribier A, Webb J, Bapat V, Reisman M, Makkar R, Leon M, Rihal C, Vahanian A, O'Neill W, Feldman T. 1-Year Outcomes of Transcatheter Mitral Valve Replacement in Patients With Severe Mitral Annular Calcification. J Am Coll Cardiol. 2018 May 1;71(17):1841-1853. doi: 10.1016/j.jacc.2018.02.054. PMID 29699609